CLINICAL TRIAL: NCT01867957
Title: A Single Blind, Randomized, Placebo Control, Phase I Study to Evaluate the Safety and Immunogenicity of the GC1109 Administered by the Intramuscular Route in Healthy Men
Brief Title: Efficacy and Safety of Anthrax Vaccine, GC1109
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry); LSK Global Pharma Services Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Myoung-don Oh, Professor, Division of Infectious Diseases, Department of Internal Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GC1109_P1_v1.2
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Anthrax
Keywords: anthrax; vaccine; bioterrorism; efficacy; safety
MeSH Terms: conditions — Anthrax | interventions — Vaccination; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Low-dose GC1109 (Experimental)
  Interventions: Biological: Low-dose GC1109
- Low-dose Placebo (Placebo Comparator)
  Interventions: Biological: Low-dose Placebo
- High-dose GC1109 (Experimental)
  Interventions: Biological: High-dose GC1109
- High-dose Placebo (Placebo Comparator)
  Interventions: Biological: High-dose Placebo

INTERVENTIONS:
Biological: Low-dose GC1109 — 50ug/dose
  Other Names: GC1109 50ug/dose (0.5 ml) vaccination
  Arms: Low-dose GC1109
Biological: High-dose GC1109 — 100ug/dose
  Other Names: GC1109 100ug/dose (1.0 ml) vaccination
  Arms: High-dose GC1109
Biological: Low-dose Placebo — 0.9% Saline 0.5 mL
  Other Names: 0.9% Saline 0.5 mL vaccination
  Arms: Low-dose Placebo
Biological: High-dose Placebo — 0.9% Saline 1.0 mL
  Other Names: 0.9% Saline 1.0 mL vaccination
  Arms: High-dose Placebo

SUMMARY:
1. BACKGROUND The newly developed anthrax vaccine GC1109 has been proven safe and effective in preclinical studies.
2. OBJECTIVE

   - To evaluate the immunogenicity and safety of the anthrax vaccine GC1109 in healthy male volunteers.
3. STUDY DESIGN

   * single-blinded
   * randomized
   * placebo controlled
   * phase 1 study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 45 years of age at the time of screening visit
2. 18.5kg/m2 ≤BMI < 30kg/m2 at the time of screening visit
3. Subjects without congenital or chronic disorder

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 0 - 28 Days

SECONDARY OUTCOMES:
Anti-protective antigen(PA) antibody level (by TNA) | Day 14, Day 28
Anti-PA Immunoglobulin G (IgG) (by ELISA) | Day 14, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea